CLINICAL TRIAL: NCT01872650
Title: A Randomized, Controlled, Clinical Trial to Assess the Effect and Safety of the C-Qur™ fiLm, an antI-adhesive Barrier for the PrevEntion of sUrgical adhesionS
Brief Title: A Trial to Assess the Effect and Safety of the C-Qur™ Film
Acronym: CLIPEUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Drs. M.W.J. Stommel, MD, University Medical Center Nijmegen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLIPEUS
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Adhesions
Keywords: postoperative adhesions; adhesion prevention; colorectal surgery; temporary ostomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No placement of an adhesion barrier
- C-Qur (Experimental): C-Qur film placement beneath the incision. Possibly placement of C-Qur film at other sites considered to be adhesiogenic (but not around the anastomosis)
  Interventions: Device: C-Qur

INTERVENTIONS:
Device: C-Qur — In subjects assigned to the treatment arm, the C-Qur™ Film must be applied beneath the incision. The C-Qur™ film can also be applied to other areas considered to be adhesiogenic (e.g. the dissection site and ostomy site but not around the anastomosis). The number of C-Qur™ Film sheets placed is limited to a maximum area of coverage of 774cm2.
  Arms: C-Qur

SUMMARY:
Adhesions develop in more than 90% of patients undergoing an intra-abdominal surgical leading to serious consequences and complications at reoperation.

The investigators initiate a prospective, randomized, controlled, multicenter trial to assess whether the use of C-Qur™ Film decreases the incidence of adhesion formation in subjects undergoing colorectal surgery. Treatment with the application of C-Qur™ Film as an adhesion prevention barrier for colorectal surgery will be compared with the control group at the second stage ostomy takedown procedure. The primary outcome evaluation will be assessment of adhesions to the incision site.

DETAILED DESCRIPTION:
Rationale:

Adhesions are fibrous bands that connect tissue surfaces where anatomical connections do not normally exist. Adhesion tenacity appears to be related to maturity, as they can be filmy or heavily vascularized with sensory nerve fibers. Adhesions are formed after a tissue surface has been injured (abrasion, desiccation, lysis, etc.) and the subsequent process of fibrinolysis is interrupted. Adhesions develop in more than 90% of patients undergoing an intra-abdominal surgical procedure. The clinically relevant symptoms of adhesion formation are small bowel obstruction, secondary infertility and pain. Other consequences and complications of postsurgical intra-abdominal adhesion formation include inadvertent enterotomy and increased dissection time due to adhesiolysis during repeat surgery. The C-Qur™ Film offers reduction of adhesion formation and the corresponding potential reductions in small bowel obstruction, secondary infertility, pain and incidence of enterotomies and prolonged dissection time during subsequent abdominal surgery.

Objective:

The primary objective is to assess whether the use of C-Qur™ Film decreases the incidence of adhesion formation in subjects undergoing colorectal surgery with a temporary loop ileostomy or loop/split colostomy. Treatment with the application of C-Qur™ Film as an adhesion prevention barrier for colorectal surgery will be compared with the control group at the second stage ostomy takedown procedure. The primary outcome evaluation will be assessment of adhesions to the incision site.

Safety objective is to assess the number and type of post-operative complications.

Study design:

This is a prospective, physician initiated, randomized, controlled, multicenter trial. Eligible subjects undergoing colorectal resection requiring temporary loop ileostomy or loop/split colostomy by laparotomy or hand assisted laparoscopy will be included in the trial. Before closure, patients are randomized 1:1 to either the treatment arm (C-Qur™ Film) or control arm (no adhesion barrier). Subjects will return 8-16 weeks post-colorectal resection to have their loop ileostomy or colostomy surgically taken down. During the loop ileostomy/colostomy takedown, adhesions will be evaluated for incidence, extent, and severity.

Study population:

Males and females 18 years of age or older, undergoing elective open or hand assisted laparoscopic colorectal resection for any colorectal disease with the formation of a temporary loop ileostomy or loop/split colostomy.

Intervention:

In subjects assigned to the treatment arm, the C-Qur™ Film must be applied under the incision. Preferably it is also applied to other areas considered to be adhesiogenic, except the anastomosis. The number of C-Qur™ Film sheets placed in the abdomen is limited to a maximum area of coverage of 774cm2 (Please refer to Table 2 in section 6.6 for the maximum number of sheets for each size).

Main study parameters/endpoints:

The primary endpoint is the incidence of adhesions to the incision site in subjects undergoing colorectal surgery with a temporary loop ileostomy or loop/split colostomy.

Secondary endpoints include:

* Incidence of adhesions to the loop ileostomy or colostomy site
* Extent and severity of adhesions to the incision site
* Extent and severity of adhesions to the loop ileostomy or colostomy sites
* Duration of ileostomy takedown from the start of the takedown to the time the bowel is repositioned in the abdomen
* Percentage (%) of abdominal wall with adhesions

Safety:

• Type and frequency of surgical and medical complications, including all types of surgical site infections

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either open or hand assisted laparoscopic colonic and/or rectal resection whereby an incision is made of 6 cm or longer
* Patients willing and capable of providing written informed consent prior to study enrolment

Exclusion Criteria:

* Pregnant women
* Patients for whom it is known, prior to the initial procedure, that loop ileostomy or colostomy closure between 8 and 16 weeks is not feasible for any reason
* Patients with known/active intra-abdominal infection such as peritonitis, abdominal abscess, anastomotic leakage or fistula (Interloop abscesses in the resection specimen is not an exclusion criterion)
* Patients with endometriosis
* Patients with known allergies to any component of the C-Qur Film device
* Patients requiring an additional procedure at the time of loop ileostomy or colostomy takedown deemed interfering with adhesion assessment by the treating surgeon.
* Patients in whom it is intended to use intraoperative lavage/irrigation with any anti-adhesion solutions other than lactated ringers and/or saline (e.g. dextran, heparin, corticosteroids, ADEPT, any other irrigant that is believed to have anti-adhesion properties ) or an adhesion barrier other than C-Qur Film™.
* Patients who have received within the last 30 days or are planned to receive systemic agents prior to the index procedure with the intention to prevent adhesion formation
* Planned chemotherapy and/or abdominal radiotherapy between index surgery and loop ileostomy or colostomy takedown
* Patients taking immune system suppressants deemed by the surgeon to interfere with wound healing (patients taking daily doses of corticosteroids exceeding 20mg within the prior 30 days are to be excluded). Patients requiring perioperative corticosteroid supplementation are not to be excluded.
* Patients with impaired immune system function or coagulation disorders deemed by the surgeon to interfere with wound healing
* Patients with a known history of severe multiple drug allergies
* Patients who have a life expectancy of less than 6 months because of a medical condition or disease state
* Any patient with a medical condition or other serious condition which will interfere with compliance and/or ability to complete this study protocol or who in the opinion of the investigator would not be a good candidate for enrolment
* Patients participating in a study of another investigational device or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
adhesions at the incision site | 8-16 weeks after index surgery
  The incidence of adhesions at the incision site

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, Study Chair — Department of Surgery, Radboud University Nijmegen Medical Center
Locations (1):
- Department of Surgery, Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Derived] Stommel MW, Strik C, ten Broek RP, van Goor H. Efficacy and safety of the C-Qur Film Adhesion Barrier for the prevention of surgical adhesions (CLIPEUS Trial): study protocol for a randomized controlled trial. Trials. 2014 Sep 26;15:378. doi: 10.1186/1745-6215-15-378. PMID 25260232